CLINICAL TRIAL: NCT00315783
Title: Comparison of Data Obtained by Echocardiography and Magnetic Resonance Imaging in Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: 2006102
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2006-04-19 (Estimated); Status verified 2006-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; echocardiography; magnetic resonance imaging
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
Compare data (structural and functional) obtained by transthoracic rest echocardiography and magnetic resonance imaging (with gadolinium) in 30 patients with hypertrophic cardiomyopathy

DETAILED DESCRIPTION:
All data from consecutive patients with HCM explored by 2D-echo or MRI in our institution will be analyzed blindly by a senior echocardiographist and a senior radiologist to highlights the respective interest of each of these examinations for the detection of structural or functional abnormalities in HCM.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic cardiomyopathy
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* Pacemaker
* IACD
* Allergy to gadolinium
* Secondary hypertrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Albert A HAGEGE, Md, PhD, Principal Investigator — Hopital Européen Georges Pompidou, Paris-FR
Locations (1):
- Hopital Européen Georges Pompidou, Paris, France